CLINICAL TRIAL: NCT00844389
Title: Near to Infrared Light Stimulation Effect on Ganglion Cell Function in Glaucomatous Optic Neuropathy
Brief Title: Near to Infrared (NIR) Light Neuroprotection in Glaucomatous Optic Neuropathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Tatiana Cevo, Universidad de Valparaíso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT45-GLAUC
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Open Angle Glaucoma
Keywords: Open Angle Glaucoma; Biophotomodulation; Near to Infrared light stimulation; Neuroprotection
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIR light (Active Comparator): Group of patients stimulated with near to infrared light daily stimulation
  Interventions: Device: Near to infrared light retinal stimulation
- Green light (Placebo Comparator): Group of patients stimulated with green light.
  Interventions: Device: Green light stimulation

INTERVENTIONS:
Device: Near to infrared light retinal stimulation — Patients will be stimulated with 660 nm light frequency through a LED device. Patients will be stimulated daily for two minutes for a 6 month period.
  Arms: NIR light
Device: Green light stimulation — Patients will be stimulated with 530 nm LED light frequency through a LED device. Patients will be stimulated daily for two minutes for a 6 month period.
  Arms: Green light

SUMMARY:
The purpose of the study is to evaluate if near-to-infrared light stimulation can improve retinal ganglion cell function in glaucomatous patients.

DETAILED DESCRIPTION:
Ganglion cell dysfunction in glaucomatous optic neuropathy has been ascribed to ganglion cell electrophysiological inactivation and to apoptotic cell death. Near-to-infrared light stimulation has been used to induce mitochondrial activation and to prevent apoptotic death through mitochondrial cytochrome oxidase c stimulation. Near-to-infrared light stimulation might be useful to induce ganglion cell activation and inhibit apoptotic cell death.

We propose that near-to-infrared light stimulation can be used as an adjuvant treatment combined with ocular hypotensive treatment in glaucomatous patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose of Ocular Hypertension (cup to disk ratio 0,6 or less, normal Humphrey 24-2 visual field with aplanatic IOP over 21 mmHg) or Mild Glaucoma (cup to disk ratio 0,6 to 0,8, characteristic Humphrey 24-2 visual field defect PSD between 3 and 6 dB).
* Visual acuity 20/40 or better

Exclusion Criteria:

* Diabetic retinopathy, Multiple Sclerosis, Parkinson disease
* Refractive error of 3 diopters or more

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Pattern electroretinogram response | Every two weeks for 4 months

SECONDARY OUTCOMES:
OCT ganglion cell layer average thickness, Visual Field defects | Every month for four months

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana E Cevo, M.D, Principal Investigator — Universidad de Valparaiso; Adrian Palacios, PhD, Study Director — Universidad de Valparaiso
Locations (1):
- Servicio de Oftalmología Hospital Van Buren, Valparaíso, Región de Valparaíso, Chile